CLINICAL TRIAL: NCT04009278
Title: Self-compression Mammography in Clinical Practice: A Randomized Clinical Trial Compared to Standard Compression Mammography
Brief Title: Self-compression Mammography in Clinical Practice
Acronym: Pristina2/TR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCT Pristina 2/TR
Record Dates: First submitted 2019-01-09; First posted 2019-07-05 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2021-01

CONDITIONS: Mammography; Breast Cancer
Keywords: Pain and discomfort
MeSH Terms: conditions — Breast Neoplasms; Pain

STUDY DESIGN:
Intervention Model Description: The study will be proposed to women presenting for a clinical mammography . Randomization will be determined by the machine's order entry system. All women will have a mammogram performed on the Pristina. In the control arm, mammography will be performed as normal clinical practice, with compression controlled by the radiographer.
  In the experimental arm the radiographer will first explain to the woman how to use the self-compression device, then position the woman's breasts and reach a compression of 5 daN, that this is a minimum but sub-optimal level of compression, and that at that point the woman will have to complete the compression to reach the optimal compression level up to an acceptable pain.
Who Masked: Outcomes Assessor
Masking Description: Each patient is identified in the study by a Subject Number (Subject No.), that is assigned when the patient is registered for mammography and is retained as the primary identifier for the patient throughout his/her entire participation in the trial.
  The allocation to experimental or control arm ill be open to patients and the research staff.
  The Image quality evaluations of Radiologists and the Radiographers are performed blindly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1. Self-compression arm (Experimental): Intervention consist in a explanation by the radiographer to the woman how to use the self-compression device, then position the woman's breasts and reach a compression of 5 daN, that this is a minimum but sub-optimal level of compression, and that at that point the woman will have to complete the compression to reach the optimal compression level up to an acceptable pain.
  Interventions: Other: Self compression arm
- 2. Control arm (No Intervention): The mammography will be performed as normal clinical practice, with compression controlled by the radiographer.

INTERVENTIONS:
Other: Self compression arm — The optimal compression level up will be under the supervision of the radiographer who will interpose the compression when a level is reached beyond which there is no further reduction in thickness (15 daN). If the woman stops at a compression of less than 10 daN and that the radiographer considers not adequate to perform a quality mammogram, the radiographer will perform the compression in conventional mode and record the passage of compression mode.
  Arms: 1. Self-compression arm

SUMMARY:
Every year millions of mammograms are performed worldwide, representing the primary examination for the early diagnosis of breast cancer. Despite continuous advances in medicine and technology, an aspect of mammography has not changed in over fifty years: the breast is still compressed on the detector because this allows to reduce the thickness of the breast thus improving the quality of the diagnostic image and reducing the dose of radiation necessary to obtain a clear image. Many women perceive as painful this compression, including women who have been treated for breast cancer.

Pain can discourage asymptomatic women to present themselves periodically to screening mammography, while an increasing number of women in follow-up after conservative surgery have to withstand the pain caused by mammography.

Some studies mention various factors that are responsible for pain when performing mammography: breast sensitivity, anxiety level, expected pain and staff attitude. Some studies have also identified breast density, breast volume and menstrual phase as other influencing factors, although not all studies support these hypothesis. The technical characteristics of the equipment can greatly affect annoyance, sense of oppression, pain. The technological proposals to reduce the discomfort of the patients concern various items: flexible compressors, self-compression devices under the supervision of the technician who performs the positioning and the minimum initial compression, environmental factors such as equipment noise reduction, chromatic, sound and sensory effects (eg: aromatic diffusers).

The aim of our study is to evaluate the effectiveness of the self-compression compared to the standard one, in reducing annoyance, a sense of oppression and pain, and to evaluate the difference of the average glandular dose given to the woman for each projection.

Self-compression may help reaching better compression tolerating the discomfort and pain induced thus allowing to achieve a lower thickness, a lower glandular dose and a better image.

ELIGIBILITY:
Inclusion Criteria:

* Women in follow-up after surgery
* Symptomatic women undergoing mammography
* Early diagnosis in asymptomatic women outside the organized screening program (these women are predominantly aged 40-44 / 75-85)
* Women with familiar risk

Exclusion Criteria:

* Augmentation prostheses
* Women in screening with active invitation
* Physical impossibility to use the self-compression command
* Inability to provide consent

Min Age: 18 Months | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Average glandular dose administered (mSv) | This outcome is measured at the baseline mammography.
  Average glandular dose administered during mammography is automatically computed by the machine according to an algorithm using the data on the quantity of radiation emitted and the radiation captured by the detector.
Image quality: radiographers' scale. | This outcome is measured at the baseline mammography.
  Radiographers evaluate the image quality after exam with a radiographer specific 3-item scale (contrast, resolution, compression) on a 0 to 5 point scale. Higher values mean better quality.
Image quality: radiologists' scale. | This outcome is measured at the baseline mammography.
  Radiologists evaluate the image quality after exam a radiologist specific 3-item scale (contrast, resolution, compression) on a 0 to 5 point scale. Higher values mean better quality.

SECONDARY OUTCOMES:
Breast thickness at the time of exposure (cm) | This outcome is measured at the baseline mammography.
  Breast thickness is measured automatically by the machine. This endpoint will be evaluated using single exposure as statistical unit, taking into account the autocorrelation of the 4 exposures in the same woman.
Maximum compression (daN) | This outcome is measured at the baseline mammography.
  Compression is measured automatically by the machine. This endpoint will be evaluated using single exposure as statistical unit, taking into account the autocorrelation of the 4 exposures in the same woman.
Pain during compression | pain will be evaluated immediately after baseline mammography execution
  visual assessment scale
Memory of pain in previous mammography | before the follow up mammography, i.e. approximately 1 year after baseline mammography
  visual assessment scale
Anxiety | Anxiety will be measured just before the baseline mammography and before the follow up mammography, i.e. approximately 1 year after baseline mammography.
  questionnaire: State Trait Anxiety Inventory for adults - form Y (D. Spielberger).
  The scale has 20 items for assessing trait anxiety and 20 for state anxiety. All items are rated on a 4-point scale. Higher scores indicate greater anxiety.
Discomfort | Discomfort will be measured just after the baseline mammography.
  Discomfort will be measured with a one-item scale with five-point range (no, slight, moderate, considerable and severe discomfort).
Execution time of the exam: | This outcome is measured at the baseline mammography.
  We evaluate: - total time (from randomization to close examination). Times are automatically registered by the radiology information system.
  - Second breast time (from the acquisition of the second right breast projection to the acquisition of the second left breast projection)
Participation in follow up mammography | 1 year (+/- 2 months) after baseline mammography
  Number of women presenting to follow up mammography (1 year +/-2 months)/number of recruited women referred to follow up mammography after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Laura Canovi, RT, Principal Investigator — Arcispedale S.Maria Nuova
Locations (1):
- Laura Canovi, Reggio Emilia, RE, Italy

IPD SHARING:
Plan to Share IPD: No
The differences in average glandular dose between the two groups will be compared with a student test if the distributions can be assimilated to a normal one and with non-parametric test in case of non-normality of the distributions.
  If the average glandular dose is not lower in the study group (superiority test) and / or the proportion of women with suboptimal compression (<10daN) and> = in the experimental group, the image quality measured with a qualitative subjective scale of the radiologist with a non-parametric test (superiority test).
  For secondary endpoints, the results will be compared between the two arms with student tests for the medium with normal distribution, non-parametric tests for non-normal distributions, while for the proportions a chi-square test will be performed.

REFERENCES:
- [Background] Miller D, Livingstone V, Herbison P. Interventions for relieving the pain and discomfort of screening mammography. Cochrane Database Syst Rev. 2008 Jan 23;2008(1):CD002942. doi: 10.1002/14651858.CD002942.pub2. PMID 18254010
- [Background] Andrews FJ. Pain during mammography: implications for breast screening programmes. Australas Radiol. 2001 May;45(2):113-7. doi: 10.1046/j.1440-1673.2001.00889.x. PMID 11380352
- [Background] Poulos A, McLean D, Rickard M, Heard R. Breast compression in mammography: how much is enough? Australas Radiol. 2003 Jun;47(2):121-6. doi: 10.1046/j.0004-8461.2003.01139.x. PMID 12780439
- [Background] Mercer CE, Hogg P, Lawson R, Diffey J, Denton ER. Practitioner compression force variability in mammography: a preliminary study. Br J Radiol. 2013 Feb;86(1022):20110596. doi: 10.1259/bjr.20110596. PMID 23385990
- [Background] Mendat CC, Mislan D, Hession-Kunz L. Patient comfort from the technologist perspective: factors to consider in mammographic imaging. Int J Womens Health. 2017 May 18;9:359-364. doi: 10.2147/IJWH.S129817. eCollection 2017. PMID 28572739
- [Background] Davey B. Pain during mammography: possible risk factors and ways to alleviate pain. Radiography. 2007;13:5
- [Background] de Groot JE, Branderhorst W, Grimbergen CA, den Heeten GJ, Broeders MJM. Towards personalized compression in mammography: a comparison study between pressure- and force-standardization. Eur J Radiol. 2015 Mar;84(3):384-391. doi: 10.1016/j.ejrad.2014.12.005. Epub 2014 Dec 13. PMID 25554008
- [Background] Feder K, Grunert JH. Is Individualizing Breast Compression during Mammography useful? - Investigations of pain indications during mammography relating to compression force and surface area of the compressed breast. Rofo. 2017 Jan;189(1):39-48. doi: 10.1055/s-0042-119450. Epub 2016 Dec 21. PMID 28002858
- [Background] Guidelines for Quality Assurance in Mammography Screening, third edition, The National Cancer Screening Service Board 2008
- [Background] de Groot JE, Broeders MJ, Grimbergen CA, den Heeten GJ. Pain-preventing strategies in mammography: an observational study of simultaneously recorded pain and breast mechanics throughout the entire breast compression cycle. BMC Womens Health. 2015;15:26. doi: 10.1186/s12905-015-0185-2. Epub 2015 Mar 15. PMID 25783657
- [Background] Van Goethem M, Mortelmans D, Bruyninckx E, Verslegers I, Biltjes I, Van Hove E, De Schepper A. Influence of the radiographer on the pain felt during mammography. Eur Radiol. 2003 Oct;13(10):2384-9. doi: 10.1007/s00330-002-1686-6. Epub 2002 Nov 14. PMID 14534806
- [Background] Lau S, Abdul Aziz YF, Ng KH. Mammographic compression in Asian women. PLoS One. 2017 Apr 18;12(4):e0175781. doi: 10.1371/journal.pone.0175781. eCollection 2017. PMID 28419125
- [Background] Taplin SH, Rutter CM, Finder C, Mandelson MT, Houn F, White E. Screening mammography: clinical image quality and the risk of interval breast cancer. AJR Am J Roentgenol. 2002 Apr;178(4):797-803. doi: 10.2214/ajr.178.4.1780797. PMID 11906848
- [Background] Shrestha S, Poulos A, The effect of verbal information on the experience of discomfort in mammography, Radiography, Volume 7, Issue 4, Pages 271-277; 2001
- [Background] Kornguth PJ, Keefe FJ, Wright KR, Delong DM. Mammography pain in women treated conservatively for breast cancer. J Pain. 2000 Winter;1(4):268-74. doi: 10.1054/jpai.2000.7884. PMID 14622609
- [Derived] Iotti V, Giorgi Rossi P, Canovi L, Guberti M, Nitrosi A, Lippolis DG, Marchesi V, Besutti G, Ottone M, Vacondio R, Pattacini P; Self-Compression Reggio Emilia Working Group. Patient-centred care with self-compression mammography in clinical practice: a randomized trial compared to standard compression. Eur Radiol. 2023 Jan;33(1):450-460. doi: 10.1007/s00330-022-09002-z. Epub 2022 Jul 22. PMID 35869315